CLINICAL TRIAL: NCT07225894
Title: Designing an Ethnodrama Addressing PrEP Stigma Toward Young Cisgender Women in Kenya
Brief Title: PrEP (Pre-exposure Prophylaxis) Stigma and Women Ethnodrama Pilot Phase
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00115054_1; R01TW012673 (NIH)
Record Dates: First submitted 2025-10-28; First posted 2025-11-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: HIV
Keywords: Stigma; HIV; PrEP
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Young women intervention cohort (Experimental): Each participant will attend all play performances in a single round (e.g., 6 plays within a week).
  Interventions: Behavioral: Ethnodrama Intervention
- Young women control cohort (No Intervention): Participants do not watch the drama performances.
- Community cohort (Experimental): This cohort consists of community members who will be identified from the audience during the first play in a round. They will be asked to watch all plays in a round.
  Interventions: Behavioral: Ethnodrama Intervention
- Audience member group (Experimental): These are audience members who heard about the play from the public announcements and chose to attend and watch the play.
  Interventions: Behavioral: Ethnodrama Intervention

INTERVENTIONS:
Behavioral: Ethnodrama Intervention — The intervention is six drama performances that are designed to transform community member beliefs about and foster support of young women's PrEP use, reduce PrEP-related enacted stigma toward young women, and reduce PrEP-related anticipated and internalized stigma among young women.
  Arms: Audience member group; Community cohort; Young women intervention cohort

SUMMARY:
The investigators will pilot test an ethnodrama intervention designed to transform community member beliefs about and foster support of young cisgender women (YCW) using Pre-exposure Prophylaxis (PrEP).

DETAILED DESCRIPTION:
In Aim 3, the investigators will pilot test the ethnodrama intervention (i.e., six plays on reducing PrEP stigma toward young women) that were pre-tested in Aim 2. The pilot evaluation will focus on evaluating logistical feasibility and describing participants' perceptions of the intervention's influence on PrEP-related stigma toward young women.

ELIGIBILITY:
Inclusion:

* Young women who are currently using or have previously used PrEP
* Community members (adult women and men) who will be identified from the audience during the first play in a round
* Adult audience members (female and male) who heard about the play from the public announcements and chose to attend and watch the play

Exclusion:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender will be self-identified
Enrollment: 160 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the drama intervention as measured by the number of plays performed as intended | Up to 1 month post-intervention
Feasibility of the drama intervention as measured by the number of study procedures implemented easily | Up to 1 month post-intervention
Feasibility of the drama intervention as measured by the estimated number of audience members | Up to 1 month post-intervention

SECONDARY OUTCOMES:
Potential effectiveness of the intervention's storylines on transforming audience members' PrEP-related perceptions as measured by a brief interviewer-administered survey using the Narrative Transportation Scale (NTS) | Immediately post-intervention
  The 12-item scale is divided into two sub-scales: engagement and personal connection. Sample items include: "I wanted to learn what happened to the women after the story ended"; "The stories in the dramas are relevant to my everyday life"; and "The stories in the drama are realistic and believable." The total score ranges from 12 to 84, where a higher score indicates greater narrative transportation.
PrEP (Pre-exposure Prophylaxis) stigma | Baseline, immediately post-intervention, and up to 3 months post-intervention
  The investigators will administer the survey at three distinct time points to assess descriptive changes in stigma-related perceptions among young women. The first administration will occur prior to the implementation of any play performances to establish baseline measures (e.g., up to several weeks prior to the first play). The second administration will take place immediately after participants have attended all six plays (e.g., up to two weeks after the last play), capturing immediate post-intervention responses. The third and final administration will occur up to three months following the last performance to assess sustained impact over time.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Corneli, PhD, MPH, Principal Investigator — Duke University
Locations (1):
- Impact Research and Development, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No